CLINICAL TRIAL: NCT01245413
Title: Controlled Randomized Study With a New Base Plate Versus SenSura Base Plate on Perspiring Skin
Brief Title: Controlled Randomized Study With Athena Base Plate Versus SenSura Base Plate on Perspiring Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Collaborators: Lægernes Test Center A/S (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CP213OC
Record Dates: First submitted 2010-11-16; First posted 2010-11-22 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Stoma; adhesive; warm; moist; cycling; men; peel-value; healthy men 50-70 years old; men with colostoma, above 18 years
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SenSura Adhesive (device) (Active Comparator): Sensura is a commercially available adhesive, that is designed to collect output from a stoma.
  Interventions: Device: SenSura
- Athena adhesive (Experimental): Athena = new test adhesive. The Athena baseplate is intended for collecting output from a stoma.
  Interventions: Device: Athena

INTERVENTIONS:
Device: SenSura — Adhesive to stoma bag
  Other Names: ostomy appliance
  Arms: SenSura Adhesive (device)
Device: Athena — Adhesive to stoma bag
  Other Names: ostomy appliance
  Arms: Athena adhesive

SUMMARY:
Aim

The aim of the Athena project is to develop an ostomy product that is softer and more flexible in order to improve the comfort for people with a stoma.

The present investigation aims at testing how well the new Athena base plate adhere to perspiring skin both with and without mechanical exposure (cycling) since the ability to adhere under normal daily activity is an important quality for Coloplast products.

Success criteria:

The investigation is an explorative investigation where the adherence of Athena on perspiring skin is evaluated. Due to the explorative nature of the study it has not been possible to define specific success criteria up front. However, the adherence qualities of Athena may not be significantly reduced compared to SenSura.

Design:

Two groups of men, one group with a colostomy and one group without a colostomy, are included. The men should be cardiovascular fit, be able to cycle for 1 hour at moderate intensity and with Athena and SenSura base plates applied on the back and stomach. The adhesion of the base plates are tested before and after the physical activities.

Population:

The population consists of two groups. Group A: Men in the age of 50-70 without a stoma who have volunteered. Group B: Men with a colostomy who have volunteered. Both groups should be cardiovascular fit (cardio investigated), and be willing to cycle for 1 hour at moderate intensity on an exercise bike.

The Athena test products are non-CE marked, non-sterile, 1-piece ostomy products with a flat custom cut base plate, a closed bag size midi or maxi with the intended use of collecting faeces from the colostomy. The comparator product is a Coloplast SenSura, 1-piece ostomy product with a closed bag. SenSura is CE-marked and launched on the market.

DETAILED DESCRIPTION:
The aim of the Athena project is to develop an ostomy product, for people with a colostomy, with better comfort than other normal ostomy products. This has been attempted through development of a soft and flexible base plate that follows the contours of the body.

It is the aim of Coloplast to gain knowledge about whether the Athena base plate can adhere to peristomal skin to the same degree as the SenSura base plate in situations of perspiration both with and without mechanical exposure.

Primary endpoint Calculation of the area of the base plate that has detached from the skin. The area is based on a visual evaluation of Athena and SenSura adhesives measured on the skin of the stomach after 1 hour of cycling at moderate intensity.

Secondary endpoint(s)

* Registration of the weight of the adhesive after physical activity on the bike and after 1 hour in a warm room.
* Evaluation of the effects on the skin measured as number of skin cells on the adhesive after use.
* Loss of liquid.
* Peel test (tractive force) of the adhesive on the skin of the stomach (mechanical exposure and perspiration).
* Peel test (tractive force) of the adhesive on the skin of the back (perspiration without the mechanical exposure).
* Calculation of the area that has detached from the skin based on a visual evaluation of the adhesives on the skin of the back (perspiration without mechanical exposure).
* Mechanical evaluation of the area of the adhesive that no longer adhere to the skin on both the stomach and on the back.

Safety endpoint(s)

* Test of health (is evaluated by the responsible physician and cardiologist).
* Test of fitness (fitness rating).
* Unexpected clinical occurrence (adverse events, AE) / Serious unexpected clinical occurrence (serious adverse events, SAE).

Criteria of success The investigation is an explorative investigation where the adherence of Athena on perspiring skin is evaluated. Due to the explorative nature of the study it has not been possible to define specific success criteria up front. However, the adherence qualities of Athena may not be significantly reduced compared to SenSura.

Design of the clinical study Study design The investigation is designed as a randomized control study with 2 groups: A and B. Group A includes 15 healthy men in the age of 50-70 years who have volunteered. Group B includes 15 men with a colostomy who have volunteered. All persons included should have a healthy cardiovascular system (see below) allowing them to accomplish one hour of cycling at moderate intensity. Both screening and test will take place at the Physicians Test Centre (Lægernes Test Center), Skodsborg Strandvej 215 A, 2942 Skodsborg, Denmark.

40 participants will be invited for screening. Those who are evaluated as suitable will be invited to proceed in the investigation. If more than 15 men without a stoma or more than 15 men with a stoma are evaluated as suitable for the test then the additional persons will be invited to register on a waiting list and they will be informed about participation in the investigation if needed. If less than 15 men without a stoma or 15 men with a stoma are evaluate as suitable then the investigation will proceed with the persons available. There will be no further recruitment of additional subjects after the screening.

The Clinical Protocol is signed by the responsible investigator at the Physicians Test Centre before the test will take place. The responsible investigator and other physicians who will act as investigators will receive thorough information about the investigation. Before recruitment of subjects the investigators will be trained in how to inform the subjects about the investigation and how to fill in the CRF (Case Report Form)(inclusive training in how to perform the different tests of adhesive qualities).

On the day of screening the subjects will be examined by an investigator with regard to health and fitness. The examination will take place at the Physicians Test Centre. The examination will also include an interview regarding life style. The cardiological data will be evaluated by a cardiologist. Persons will be invited for another one or two test days if the investigator finds that the person is able to do one hour of cycling at moderate intensity without risk and otherwise comply with the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Group A: Men without a stoma in the age of 50-70 years Group B: Men with a stoma

Inclusion criteria:

To be included in the investigation, the subjects in Group A must comply with the following selection criteria:

* Have signed informed consent and letter of attorney
* Be a man in the age of 50-70 years
* Is capable of understanding the experiment
* Have a BMI (body mass index) between 20-30 kg/m2
* Is willing to test the adhesives from the two Coloplast products, Athena and SenSura
* Is evaluated as suitable for inclusion according to cardiovascular test and fitness test performed at the screening

To be included in the investigation, the subjects in Group B must comply with the following selection criteria:

* Have signed informed consent and letter of attorney
* Be a man of at least 18 years of age
* Have a colostomy with a max width of 45 mm and have had the colostomy for at least 3 months
* Is capable of understanding the experiment
* Have a BMI between 20-30 kg/m2
* Is willing to test the adhesives from the two Coloplast products, Athena and SenSura
* Is evaluated as suitable for inclusion according to cardiovascular test and fitness test performed at the screening

Exclusion Criteria:

* Subjects who comply with the following criteria must be excluded from the investigation:

  * Have dermatological problems
  * Currently receiving or have within the past 2 months received radio- and/or chemotherapy.
  * Have elevated cholesterol levels, elevated blood pressure, diabetes or any form of cardiovascular disease.
  * Currently receiving or have within the last 3 weeks received local treatment with steroids (ointment or creme) on back or stomach*
  * Group A may not have a stoma
  * Group B may not use convex base plates * Radio- and chemotherapy can lead to changes in the skin and intestine. It is known that steroid can lead to fragile skin which can affect application and removal of the adhesive

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Hyldahl, MD, Principal Investigator — Lægehuset
Locations (1):
- Lægernes Test Center A/S, Skodsborg, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 healthy volunteers and 12 colostomists were recruited to the study. The colostomist were recruited from a user data base in Denmark. The healthy volunteers were recruited by advertising in local news papers, on www.forsøgsperson.dk and by poster at"Skodsborg hotel og spa" (a fitness centre)
Pre-assignment Details: 32 subjects were enrolled and randomised in the study.
Groups:
- SenSura Adhesive: Sensura is an already commercially available baseplate. Designed to collect output from a stoma(e.g an ileostomy and colostomy).
- Athena Adhesive: Athena =the new test product. The Athena in this trails is an adhesive. The intend use is collecting output from a stoma (e.g an ileostomy and colostomy).
Period: Sensura First,
Arm/Group | SenSura Adhesive | Athena Adhesive
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Athena First,
Arm/Group | SenSura Adhesive | Athena Adhesive
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Entire study population = all participlants enrolled in the study
Arm/Group | Entire Study Population
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 63.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Visual Inspection of Baseplate Loosening
Description: The area of the adhesive that was detached from the skin based on visual evaluation of the Athena and Sensura adhesives on the stomach after 1 hour of cycling at moderate intensity. The evaluation was done by marking the detached areas at the baseplate on a transparent wound tracing sheet with a permanent marker. Subsequently the areas were measured by scanning the tracing sheet and calculating the area with the use of Imagepro image macro which calculates the result in cm^2
Time Frame: 1 hour
Population: ITT
Measure: Mean (Standard Deviation); unit: cm^2
Groups:
- SenSura Adhesive: Reference adhesive which is commercially available.
- Athena Adhesive: New test adhesive
Arm/Group | SenSura Adhesive | Athena Adhesive
Number analyzed (Participants) | 32 | 32
cm^2 | 3.77 (5.48) | 4.88 (4.95)

ADVERSE EVENTS:
Groups:
- SenSura Adhesive; Athena Adhesive: base-plate adhesion to skin
Arm/Group | SenSura Adhesive | Athena Adhesive
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days